CLINICAL TRIAL: NCT01640678
Title: Autologous Cell Suspension Grafting Using ReCell in Vitiligo and Piebaldism Patients: a Randomized Controlled Pilot Study
Brief Title: Autologous Cell Suspension Grafting Using ReCell in Vitiligo and Piebaldism Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Lisa Komen, Drs., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: METC2012_052
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Piebaldism; Segmental Vitiligo
MeSH Terms: conditions — Piebaldism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ReCell epidermal cell suspension grafting (Experimental): CO2 laser abrasion + ReCell epidermal cell suspension + UV-therapy
  Interventions: Procedure: ReCell epidermal cell suspension grafting
- CO2 laser abrasion + UV-therapy (Active Comparator): According to current standard of care procedures the treatment site will be superficially abraded using an ablative laser (10,600nm CO2 laser)
  Interventions: Procedure: CO2 laser abrasion + UV-therapy
- No treatment + UV-therapy (No Intervention)

INTERVENTIONS:
Procedure: ReCell epidermal cell suspension grafting — According to current standard of care procedures the treatment site will be superficially abraded using an ablative laser (10,600nm CO2 laser) after which the prepared ReCell cell suspension will be sprayed on.
  Arms: ReCell epidermal cell suspension grafting
Procedure: CO2 laser abrasion + UV-therapy — According to current standard of care procedures the treatment site will be superficially abraded using an ablative laser (10,600nm CO2 laser)
  Arms: CO2 laser abrasion + UV-therapy

SUMMARY:
Autologous epidermal cell suspension grafting is an effective method of surgical treatment in vitiligo, which is suitable for treating larger areas with better cosmetic results as compared to other grafting methods. The ReCell Autologous Cell Harvesting Device (Avita Medical Europe Limited, Cambridge, UK) is an autologous cell harvesting device which, compared to other forms of autologous epidermal cell suspension grafting, is easier in use showing similar results. Furthermore, the ReCell device needs no laboratory facilities. Therefore, it is promising for patients with large vitiligo and piebaldism lesions.

Objectives: Primary: to asses the efficacy and safety of autologous epidermal cell suspension grafting with the ReCell device after CO2 laser abrasion compared to CO2 laser abrasion alone and no treatment, in patients with piebaldism and stable vitiligo. Secondary: to assess the practical aspects and patients satisfaction of autologous epidermal cell suspension grafting with the ReCell device.

Study design: Prospective observer blinded randomized controlled pilot study. Study population: 10 patients ≥ 18 years with stable segmental vitiligo or piebaldism who are under treatment at the Netherlands Institute for Pigment Disorders (NIPD) at the Academic Medical Centre University of Amsterdam.

Methods: Three depigmented regions on the trunk or proximal extremities will be randomly allocated to; CO2 laser abrasion + ReCell autologous cell suspension grafting, or CO2 laser abrasion, or no treatment. After the transplantation, UV-treatment according to the standard treatment protocol of the NIPD will be started on all sites and continued for 3 months. Three and six months after grafting, the percentage of repigmentation of the lesions will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* patient with piebaldism
* Patients with segmental vitiligo,stable since 12 months without systemic therapy or topical therapy as defined by the absence of new lesions and/or enlargement of existing lesions
* with at least three depigmented skin lesions on the proximal extremities or trunk larger than 3x3 cm or one lesion of at least 9x3 cm
* Age >18
* willing and able to give written informed consent

Exclusion Criteria:

* UV therapy or systemic immunosuppressive treatment during the last 12 months
* Local treatment of vitiligo during the last 12 months
* Vitiligo lesions with follicular or non-follicular repigmentation
* Skin type I
* Recurrent HSV skin infections
* Hypertrophic scars
* Keloid
* Cardial insufficiency
* Patients with a history of hypersensitivity to (UVB or UVA) light and/or allergy to local anesthesia.
* Patients who are pregnant or breast-feeding
* Patients not competent to understand the procedures involved
* Patients with atypical nevi
* Patients with a personal history of melanoma or non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
degree of repigmentation | 6 months
  Objective assessment of the degree of repigmentation 6 months after autologous epidermal cell suspension grafting. Assessment will be done by standardized photographs and a digital image analysis system.

SECONDARY OUTCOMES:
Visual assessment of side effects per treatment region | 6 months
  Visual assessment of side effects per treatment region (hyper pigmentation, hypo pigmentation and scar on a scale from 0-3) will be done by a blinded investigator
General outcome assessed by the patient | 6 months
  General outcome will be assessed by the patient per treatment region on a scale from 0-3 (Poor, Moderate, Good, and Excellent)

CONTACTS AND LOCATIONS:
Locations (1):
- The Netherlands Institute for pigment disorders, AMC, Amsterdam, Netherlands